

# **Non-Interventional Study (NIS) Protocol**

| Document Number: | c39084239-01 |
|---|---|
| BI Study Number: | 1199-0471 |
| BI Investigational Product(s): | Nintedanib |
| Title: | Real-World Medication Adherence Trajectories to Nintedanib among<br>Idiopathic Pulmonary Fibrosis Patients |
| Brief lay title: | Adherence to Nintedanib among IPF Patients |
| Protocol version identifier: | 1.0 |
| Date of last version of protocol: | Not applicable |
| PASS: | No |
| EU PAS register number: | Will be registered |
| Active substance: | Not applicable |
| Medicinal product: | Nintedanib (Ofev) |
| Product reference: | Not applicable |
| Procedure number: | Not applicable |
| Marketing authorisation holder(s): | Not applicable |
| Joint PASS: | No |
| Research question and objectives: | <ol> <li>Identification of adherence patterns of nintedanib among idiopathic pulmonary fibrosis (IPF) patients.</li> <li>Understanding characteristics of patients within each nintedanib adherence trajectory among IPF patients.</li> </ol> |
| Country(-ies) of study: | United States |
| Author: | |

# Boehringer Ingelheim Non-Interventional Study (NIS) Protocol BI Study Number 1199-0471

**Page 2 of 42** 

c39084239-01

| Marketing authorisation holder(s): | NA NA |
|---|---|
| Date: | 12 May 2022 |
| Page 1 of 42 | |
| Proprietary confidential information © 2022 Boehringer Ingelheim Group of companies. All rights reserved. This document may not - in full or in part - be passed on, reproduced, published or otherwise used without prior written permission | |

# 1. TABLE OF CONTENTS

| TIT | `LE PAGE | | 1 |
|-----|-----------|-------------------------------------|-----|
| 1. | TABLE O | F CONTENTS | 3 |
| 2. | LIST OF A | ABBREVIATIONS | 5 |
| 3. | RESPONS | SIBLE PARTIES | 6 |
| 4. | ABSTRAG | CT | 7 |
| 5. | AMENDM | MENTS AND UPDATES | .10 |
| 6. | MILESTO | NES | .11 |
| 7. | RATIONA | ALE AND BACKGROUND | .12 |
| 8. | RESEARC | CH QUESTION AND OBJECTIVES | .14 |
| 9. | RESEARC | CH METHODS | .15 |
| 9 | 0.1 | STUDY DESIGN | .15 |
| 9 | 0.2 | SETTING | .16 |
| | 9.2.1 | Study sites | .16 |
| | 9.2.2 | Study population | .16 |
| | 9.2.3 | Study visits | .17 |
| | 9.2.4 | Study discontinuation | .17 |
| 9 | 0.3 | VARIABLES | .17 |
| | 9.3.1 | Exposures | .17 |
| | 9.3.2 | Outcomes | .17 |
| | 9.3.2.1 | Primary outcomes | .17 |
| | 9.3.3 | Covariates | .18 |
| 9 | 0.4 | DATA SOURCES | .25 |
| 9 | 0.5 | STUDY SIZE | .25 |
| 9 | 0.6 | DATA MANAGEMENT | .26 |
| 9 | 0.7 | DATA ANALYSIS | .26 |
| | 9.7.1 | Main analysis | |
| | 9.7.2 | Additional analysis | .27 |
| 9 | 0.8 | QUALITY CONTROL | |
| 9 | 0.9 | LIMITATIONS OF THE RESEARCH METHODS | .28 |
| 9 | 2.10 | OTHER ASPECTS | .29 |
| | 9.10.1 | Data quality assurance | .29 |

| Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its | arrinated companies |
|---|---|

| | 9.10.2 | Study records | 29 |
|---|---|---|---|
| 10. | PROTE | CTION OF HUMAN SUBJECTS | 30 |
| | ).1<br>ONSENT | STUDY APPROVAL, PATIENT INFORMATION, AND INFORMED | .30 |
| 10 | ).2 | STATEMENT OF CONFIDENTIALITY | 30 |
| 11.<br>REA | | GEMENT AND REPORTING OF ADVERSE EVENTS/ADVERSE | .31 |
| | l.1<br>ND REPOF | ADVERSE EVENT AND SERIOUS ADVERSE EVENT COLLECTION | |
| 12. | PLANS | FOR DISSEMINATING AND COMMUNICATING STUDY RESULTS . | 32 |
| 13. | REFERI | ENCES | 33 |
| 13 | 3.1 | PUBLISHED REFERENCES | 33 |
| 14. | ANNEX | TURES | 37 |
| A | NNEX 1. L | IST OF STAND-ALONE DOCUMENTS | 38 |
| A | NNEX 2. E | NCEPP CHECKLIST FOR STUDY PROTOCOLS | 39 |
| A. | NNEX 3. A | DDITIONAL INFORMATION | 40 |
| A <sup>-</sup> | NNEX 4. R | EVIEWERS AND APPROVAL SIGNATURES | 41 |

## 2. LIST OF ABBREVIATIONS

ADR Adverse Drug Reaction

AE Adverse Event

AESI Adverse Event of Special interest

CA Competent Authority
CCDS Company Core Data Sheet
CI Confidence Interval
CML Local Clinical Monitor

CRA Clinical Research Associate

CRF Case Report Form

CTCAE Common Terminology Criteria for Adverse Events

CTP Clinical Trial Protocol

eCRF Electronic Case Report Form

ENCePP European Network of Centres for Pharmacoepidemiology and

Pharmacovigilance

FDA Food and Drug Administration
GBTM Group-Based Trajectory Model

GCP Good Clinical Practice

GEP Good Epidemiological Practice

GPP Good Pharmacoepidemiology Practice GVP Good Pharmacovigilance Practices

IB Investigator's Brochure

IECIndependent Ethics CommitteeIPFIdiopathic Pulmonary FibrosisIRBInstitutional Review BoardMAHMarketing Authorization Holder

MedDRA Medical Dictionary for Regulatory Activities

NIS Non-Interventional Study

OOP Out Of Pocket

PASS Post-Authorization Safety Study PDC Proportions of Days Covered SAE Serious Adverse Event

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 3. RESPONSIBLE PARTIES

| BI NIS |
|--------|

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 4. ABSTRACT

| Name of company | y: | | |
|---|---|---|---|
| Boehringer Ingelheim | | | |
| Name of finished<br>product:<br>Nintedanib (Ofev) | medicinal | | |
| Name of active in<br>Nintedanib (Ofev) | 0 | | |
| Protocol date: | Study<br>number: | Version/Revision: | Version/Revision date: |
| 12 May 2022 | 1199-0471 | 1.0 | NA |
| Title of study: | | edication Adherence Trajec<br>nonary Fibrosis Patients | tories of Nintedanib among |
| Rationale and background: | Medication adherence is of great importance to health care stakeholders. The most common method to measure adherence in real-world settings is via the proportion of days covered (PDC) in prescription drug claims databases. However, PDC is limited by its inability to distinguish between different patterns of adherence over time. This study will use group-based trajectory modeling (GBTM) to assess adherence trajectories to nintedanib and patient characteristics associated with those trajectories. The results of this study can help providers/payers to better identify adults with IPF who are at high risk of nintedanib non-adherence. The identified non-adherence trajectories may highlight the need for a targeted intervention strategy to improve adherence in patients with each trajectory. | | |
| Research question and objectives: | Identification of adherence trajectories of nintedanib use among IPF patients. Understanding characteristics of patients within each nintedanib adherence trajectory among IPF patients. | | |
| Study design: | This is a non-interventional, retrospective cohort study. | | |

| Name of compan | y: | | |
|---|---|---|---|
| Boehringer Ingelh | eim | | |
| Name of finished<br>product:<br>Nintedanib (Ofev) | | | |
| Name of active in<br>Nintedanib (Ofev) | 0 | | |
| Protocol date: | Study<br>number: | Version/Revision: | Version/Revision date: |
| 12 May 2022 | 1199-0471 | 1.0 | NA |
| Population: | | ole will consist of community in the IPF who initiate treat | • |
| Variables: | The main study outcome is nintedanib adherence trajectories. A range of predictor variables will be measured in the administrative data during the baseline and index date, including patient demographic characteristics (e.g., age, sex, race/ethnicity), Social Deprivation Index, residential location, clinical characteristics (e.g., comorbidity index, IPF-related costs and use), and all-cause health care costs and use. | | |
| Data sources: | This study will use administrative enrollment and claims data from the U.S. federal Medicare program for beneficiaries aged 65 years and older who were continuously enrolled in Original Medicare insurance coverage, including Parts A, B and D. The study will use Medicare data covering the period from October 1, 2013 through December 31, 2019. | | |
| Study size: | The minimum needed sample size for GBTM analysis is 500. A prior study found 1,464 Medicare beneficiaries who initiated nintedanib between 10/15/2014 and 12/31/2015 (Corral, Chang et al., 2020). By covering a longer period with the same data, this study should have sufficient sample. | | |
| Data analysis: | In the first part, monthly trends in nintedanib PDC will be analysed via GBTM estimation, which assumes there is a fixed number of latent clusters of individuals who share a common outcome pattern. The methodology will yield estimated probabilities of cluster membership for each individual and an estimated trajectory curve over time for each cluster. In the second part, multinomial logistic models will be estimated to identify individual-level predictors of cluster membership. | | |
| Milestones: | The analytic database is expected to be constructed by August 30, 2021, pending access to the Medicare data. Data analyses are expected to be completed by October 15, 2021. A draft report of the findings from this study is expected to be available for review by November 15, 2021 and | | |

| Name of company: | | | |
|---|---|---|---|
| Boehringer Ingelhei | im | | |
| Name of finished medicinal product: Nintedanib (Ofev) | | | |
| Name of active ing<br>Nintedanib (Ofev) | redient: | | |
| Protocol date: Study number: | | Version/Revision: | Version/Revision date: |
| 12 May 2022 | 1199-0471 | 1.0 | NA |
| | completed by Fe | bruary 15, 2022. | |

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 5. AMENDMENTS AND UPDATES

None.

# 6. MILESTONES

| Milestone | Date |
|-----------------------------------|----------|
| First draft of synopsis | 2/1/21 |
| VDT synopsis review | 2/25/21 |
| IET synopsis review | 4/23/21 |
| Kick-off meeting with vendor | 05/07/21 |
| NPCC synopsis review | 05/21/21 |
| Study protocol first draft | 06/01/21 |
| Study protocol VDT and NIS review | 07/22/21 |
| Study protocol NPCC review | 08/17/21 |
| Study protocol final draft | 08/20/21 |
| Analytical database creation | 08/30/21 |
| Descriptive results to BI | 09/15/21 |
| GBTM results to BI | 10/15/21 |
| Final report first draft | 11/15/21 |
| Final report comments from BI | 01/15/22 |
| Final report final draft | 02/15/22 |

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 7. RATIONALE AND BACKGROUND

Medication adherence is of great importance to health care stakeholders based on increasing evidence of prevalence of non-adherence to chronic medications in the United States (Desai et al., 2019) and increasing evidence that adherence is associated with better health outcomes and lower costs (Cutler et al., 2018). There are several ways by which adherence to medications can be measured. Each of these methods has its own strengths and limitations (Forbes et al., 2018). Direct methods, which include blood drug assays, and direct observation of the patients are expensive, laborious, and time intensive (Farmer, 1999). In real-world settings, use of prescription claims databases, patient self-report, pill counts, and electronic monitoring are the common measures of adherence (Lam and Fresco, 2015). The most common method to measure adherence in real-world settings is via the proportion of days covered (PDC) in prescription drug claims databases (Harbaugh and Cooper, 2018). PDC has been defined as the number of days supplied of a specific medication in the follow-up period divided by the total number of days during follow-up, multiplied by 100 to yield a percentage from 0%–100% (Raebel et al., 2013).

Although PDC is useful in that it offers in a single number a metric of medication adherence over a predefined period of time, it is also limited because it does not distinguish between different patterns of adherence over that same period (Alhazami et al., 2020). For example, a patient who took medications every other day for a year would have a PDC of 50%; likewise, a patient who took the medication for the first 6 months uninterrupted and then not again for the remainder of the year would also have a PDC of 50%. Distinguishing these different patterns is critical to understanding adherence to prescription medication and designing interventions to improve adherence.

One alternative is to detect trajectories of adherence over time across patients using group-based trajectory modeling (GBTM) (Nagin and Odgers, 2010). GBTM has been applied with increasing frequency for this purpose in several conditions (Alhazami et al., 2020; Bateman et al., 2016; Dillon et al., 2018; Feldman et al., 2018; Franklin et al., 2018; Franklin et al., 2018; Franklin et al., 2015; Franklin et al., 2013; Hargrove et al., 2017; Juarez et al., 2015; Kim et al., 2017; Li et al., 2014; Lo-Ciganic et al., 2016; MacEwen et al., 2016; Paranjpe et al., 2020; Vadhariya et al., 2019; Wang et al., 2019; Zongo et al., 2019). In most of these studies, monthly PDC was assessed for each patient, and a GBTM was fit on the patient-level sequences of monthly PDC values to identify a best-fitting set of adherence trajectories as well as, for each patient, estimates of the probability of belonging to each trajectory group.

Studies that examine adherence trajectories with GBTMs frequently include analyses of the predictors of patients' membership in trajectory groups. Individual characteristics that have been observed to be related to adherence trajectories include age, race, sex, disease severity, comorbidity burden, educational attainment, and socioeconomic status (Alhazami et al., 2020).

Adherence to nintedanib has been evaluated in a few recent studies in the United States. Recent observational studies of nintedanib and pirfenidone suggest that despite different side-

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

effect profiles, adherence to and persistence with therapy are similar. Adherence (measured as PDC  $\geq$  80%) of nintedanib during one year has been estimated at 60.5% (<u>Corral, Chang, et al., 2020</u>), 51% (<u>Corral, DeYoung, and Kong, 2020</u>), and 71.3% (<u>Ipatova et al., 2019</u>). No studies to our knowledge have analyzed nintedanib adherence using GBTM or comparable methods nor have any studies assessed predictors of adherence.

Therefore, the objective of this study is to assess nintedanib adherence trajectories using GBTMs and understand characteristics of patients within each trajectory. The results of this study can help providers and payers to better identify adults with IPF who are at high risk of nintedanib non-adherence. The identified non-adherence trajectories may highlight the need for a fit-for-targeted intervention strategy to improve adherence in patients within each trajectory.

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 8. RESEARCH QUESTION AND OBJECTIVES

This study has two objectives:

- 1. Identification of adherence trajectories of nintedanib among IPF patients.
- 2. Understanding characteristics of patients within each nintedanib adherence trajectory among IPF patients.

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 9. RESEARCH METHODS

## 9.1 STUDY DESIGN

This is a non-interventional cohort study using existing administrative data from the U.S. Medicare program. There will be no comparison groups nor any exposure variables. As shown in Figure 1, the study sample will consist of community-dwelling Medicare beneficiaries with IPF who initiated treatment with nintedanib between 10/01/2014 to 12/31/2018. To allow for a one-year baseline period and one-year follow-up period for all beneficiaries who initiated nintedanib between 10/01/2014 and 12/31/2018, the span of data will be from 10/01/2013 to 12/31/2019.



Figure 1 Study design schematic

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 9.2 SETTING

#### 9.2.1 Study sites

The study will use 100% Medicare claims and enrollment data from the U.S. Medicare program on community-dwelling beneficiaries continuously enrolled in traditional, or fee-for-service, Medicare insurance coverage for inpatient hospital, skilled nursing and outpatient facility services (Part A), physician and other professional services (Part B), and outpatient prescription drugs (Part D).

The enrollment file contains monthly information on individuals' enrollment in each part of Medicare, demographic information, residential location (at the 5-digit ZIP Code level), and date of death.

Claims data are available for all medical services covered by the program and are organized into data files based on the nature and source of the claim. The Inpatient, Outpatient, and SNF files include institutional claims from hospitals for inpatient and outpatient services and from nursing homes for short-stay "skilled" admissions, respectively. The Carrier file includes fee-for-service claims submitted by professional providers, including physicians, physician assistants, clinical social workers, nurse practitioners. (Claims for some organizational providers, such as free-standing facilities are also found in the Carrier file. Examples include independent clinical laboratories, ambulance providers, free-standing ambulatory surgical centers, and free-standing radiology centers.) Separate files include claims for durable medical equipment, home health visits and hospice care.

Pharmacy Part D claims include complete prescription drug information, and all standardized prescription-level fields collected on a typical pharmacy claim (e.g., date of fill or refill, drug name and class, strength, quantity, and days' supply).

## 9.2.2 Study population

Inclusion criteria:

- Newly initiated nintedanib during 10/01/2014 to 12/31/2018 (see tab "T1 ANTIFIB RX" in standalone document "Code List.xlsx")
- Were at least 66 years old as of the date of their first nintedanib prescription claim (index date)
- Qualified for Medicare based on age
- Had at least 12 months of continuous enrollment in Medicare Parts A, B and D before (baseline period) and 12 months after the index date (follow-up period)
- Had at least one inpatient or two outpatient claims (≥14 days apart) with a diagnosis code for IPF (ICD-10-CM: J84.112; ICD-9-CM: 516.31) during the baseline period (see tab "T3 IPF DX" in standalone document "Code List.xlsx

# Non-Interventional Study (NIS) Protocol

## **BI Study Number 1199-0471**

c39084239-01

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### Exclusion criteria:

- Had any history of pirfenidone or nintedanib use during the baseline period (see tab "T1 ANTIFIB RX" in standalone document "Code List.xlsx")
- Had any history of lung transplant during the baseline, index date or follow-up periods (see tabs "T4 LUNG\_TRANS PR" and "T5 LUNG\_TRANS DX" in standalone document "Code List.xlsx")
- Had any claims for skilled nursing facility, long-term care facility or hospice during the baseline, index date or follow-up period
- Had evidence (≥2 ICD-9-CM or ICD-10-CM diagnosis codes on different dates)
  during the baseline period of any of the following conditions: lung cancer,
  autoimmune, or connective tissue diseases (i.e. rheumatoid arthritis (RA), sarcoidosis,
  systemic lupus erythematosus (SLE), dermatopolymyositis, systemic sclerosis,
  Sjogren's, and mixed connective tissue disease (CTD)) during the baseline period
  (Appendix-1)
- Had dual eligibility of Medicare and Medicaid.
- Had history of using pirfenidone at the same time with nintedanib during follow-up

#### 9.2.3 Study visits

Not applicable.

#### 9.2.4 Study discontinuation

Not applicable

#### 9.3 VARIABLES

## 9.3.1 Exposures

This is a study of nintedanib adherence patterns, and all the included patients will be patients with a prescription claim for nintedanib.

#### 9.3.2 Outcomes

#### 9.3.2.1 Primary outcomes

The main outcome of this study is adherence trajectories to nintedanib. This study will use the GBTM method to identify trajectories of adherence.

For this purpose, first claim for nintedanib will be identified in the Part D claims file based on the presence of an 11-digit NDC code for nintedanib (00597-0143-60, 00597-0145-60 [CanMED, 2021]). Nintedanib supply calendars will be constructed for the all twelve 30-day time intervals following the individual's nintedanib initiation date based on each claim's service date and days' supply.

-Supply will be assigned as 1 for each day with positive days' supply of nintedanib.

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

- -If a patient has multiple prescription claims for nintedanib on the same date, the maximum of days' supply will be calculated across the claims and applied to the supply calendar.
- -Stockpiling will be implemented if a patient has prescription claims for nintedanib that overlap. Days' supply for the newer claim will be postponed to the first day after end of the older claim's supply.
- -For each 30-day month following the nintedanib initiation date, PDC will be calculated as the sum of days with supply divided by 30.

In this way, we are able to calculate monthly nintedanib proportion of days covered. By using the twelve 30-days PDC values as outcomes in the GBTM, the probabilities that a given individual is in each of the latent clusters will be calculated by the GBTM estimation procedure. GBTMs will be estimated using the Stata plugin traj (Jones and Nagin, 2013).

#### 9.3.3 Covariates

The index date will be defined as the date of the beneficiary's first Part D claim for nintedanib. The baseline period will consist of the 360 consecutive days ending the day before the index date. The follow-up period will consist of the 360 consecutive days starting with the index date.

| Variable | Description |
|---|---|
| Demographic and socioeconomic characteristics | |
| Age | Age as of index date in years rounded to the nearest whole number will be calculated based on the difference between the beneficiary's birth date and index date. |
| Age group | Age group will be a categorical variable for age defined as one of 65–74, 75–84, 85+. |
| Female | Female will be a binary indicator for whether the beneficiary was female as indicated on the enrollment record covering the index date. |
| Race | Race will be a categorical variable for the beneficiary's self-reported race/ethnicity taking the categories Non-Hispanic White, Black or African-American, Other, Asian/Pacific Islander, Hispanic, American Indian/Alaska Native, and unknown race from the enrollment record covering the index date. |
| Census region | Census region will be a categorical variable defined by categorizing the beneficiary's state of residence into Census regions (Northeast, South, Midwest, West) from the enrollment record covering the index date (see tab "T2 STATES" in |

| Variable | Description |
|---|---|
| | standalone document "Code_List.xlsx"). |
| Index year | Index year will be a categorical variable defined as the year of the index date and will take the values, 2014, 2015, 2016, 2017 or 2018. |
| Social deprivation index | Social deprivation index will be a continuous variable ranging between 0 and 100 representing the Social Deprivation Index for the beneficiary's residential ZIP Code as calculated by the Social Deprivation Index "is a composite measure of seven demographic characteristics collected in the American Community Survey (ACS): percent living in poverty, percent with less than 12 years of education, percent single parent household, percent living in rented housing unit, percent living in overcrowded housing unit, percent of households without a car, and percent non-employed adults under 65 years of age." This version was calculated in 2015 using data from 2015 and updates the original version created by Butler et al. (2013). Higher values for the Social Deprivation Index indicate more social deprivation. |
| Clinical characteristics | |
| Combined comorbidity index | The combined comorbidity index will be a continuous comorbidity score ranging from 0 to 26 as measured from comorbidity diagnosis codes in any position on inpatient, outpatient and Carrier claims that occurred during the baseline period. The combined comorbidity score is based on research by Gagne et al. (2011) and Sun et al. (2017) to identify the conditions in the union of the two most-popular comorbidity indexes used in administrative claims data, the Charlson index and the Elixhauser index. For a sample of Medicare beneficiaries, Gagne et al. (2011) found that a subset of 20 conditions predicted mortality at 30, 60, 90 and 180 days, and 1 year more accurately than either of the two indexes on their own. Moreover, unlike the Charlson and Elixhauser indexes, Gagne et al.'s (2011) combined index is not conditioned on inpatient hospital admission. |

| Variable | Description |
|---|---|
| | The 20 conditions in <u>Gagne et al.'s (2011)</u> combined comorbidity index (with their weights in parentheses) include: |
| | - Metastatic cancer (5), |
| | - Congestive heart failure (2), |
| | - Dementia (2), |
| | - Renal failure (2), |
| | - Weight loss (2), |
| | - Hemiplegia (1), |
| | - Alcohol abuse (1), |
| | - Any tumor (1), |
| | - Cardiac arrhythmias (1), |
| | - Chronic pulmonary disease (1), |
| | - Coagulopathy (1), |
| | - Complicated diabetes (1), |
| | - Deficiency anemia (1), |
| | - Fluid and electrolyte disorders (1), |
| | - Liver disease (1), |
| | - Peripheral vascular disease (1), |
| | - Psychosis (1), |
| | - Pulmonary circulation disorders (1), |
| | - HIV/AIDS (-1), and |
| | - Hypertension (-1). |
| Pulmonary hypertension | A binary indicator for whether the beneficiary had a diagnosis code for pulmonary hypertension on at least one inpatient, outpatient or Carrier claim that occurred during the baseline period (see tab "T7 PULM_HTN DX" in standalone document "Code_List.xlsx"). |
| Gastroesophageal reflux | A binary indicator for whether the beneficiary had a diagnosis code for gastroesophageal reflux disease on at least one inpatient, outpatient or Carrier claim that occurred during the baseline period (see tab "T8 GASTR_REFLX DX" in standalone document "Code_List.xlsx"). |
| Asthma | A binary indicator for whether the beneficiary had |

| Variable | Description |
|---|---|
| | a diagnosis code for asthma on at least one inpatient, outpatient or Carrier claim that occurred during the baseline period (see tab "T9 ASTHMA DX" in standalone document "Code_List.xlsx"). |
| Sleep apnea | A binary indicator for whether the beneficiary had a diagnosis code for obstructive sleep apnea on at least one inpatient, outpatient or Carrier claim that occurred during the baseline period (see tab "T10 SLEEP_APNEA DX" in standalone document "Code_List.xlsx"). |
| Lung biopsy | A binary indicator for whether the beneficiary had a diagnosis or procedure code for a lung biopsy on at least one inpatient, outpatient or Carrier claim that occurred during the baseline period (see tab "T11 LUNG_BIOPSY PR" in standalone document "Code_List.xlsx"). |
| HRCT scan | A binary indicator for whether the beneficiary had a procedure code for a high-resolution computerized tomography scan on at least one inpatient, outpatient or Carrier claim that occurred during the baseline period (see tab "T12 HRCT_SCAN PR" in standalone document "Code_List.xlsx"). |
| Oxygen | A binary indicator for whether the beneficiary had a diagnosis, procedure revenue center code for oxygen therapy or supplemental oxygen on at least one inpatient, outpatient, Carrier, skilled nursing facility, home health or durable medical equipment claim that occurred during the baseline period (see tabs "T13 OXYGEN PR", "T14 OXYGEN REV" and "T15 OXYGEN DX" in standalone document "Code_List.xlsx"). |
| Pulmonary rehabilitation | A binary indicator for whether the beneficiary had a procedure or revenue center code for pulmonary rehabilitation services on at least one inpatient, outpatient, Carrier, skilled nursing facility, home health or durable medical equipment claim that occurred during the baseline period (see tabs "T16 PULM_REHAB PR" and "T17 PULM_REHAB REV" in standalone document "Code_List.xlsx"). |
| Ventilator use | A binary indicator for whether the beneficiary had a |

| Variable | Description |
|---|---|
| | diagnosis or procedure code for ventilator use on at least one inpatient, outpatient or Carrier claim that occurred during the baseline period (see tabs "T18 VENT_USE PR" and "T19 VENT_USE DX" in standalone document "Code_List.xlsx"). |
| COPD | A binary indicator for whether the beneficiary had a diagnosis code for chronic obstructive pulmonary disease on at least one inpatient, outpatient or Carrier claim that occurred during the baseline period (see tab "T20 COPD DX" in standalone document "Code_List.xlsx"). |
| Hypoxia | A binary indicator for whether the beneficiary had a diagnosis code for hypoxia on at least one inpatient, outpatient or Carrier claim that occurred during the baseline period (see tab "T21 HYPOXIA DX" in standalone document "Code_List.xlsx"). |
| Pharmacy use and spending | |
| Medication count | The count of the number of unique outpatient prescription medications for which beneficiary has Part D claims during the baseline period |
| Total pharmacy spending | A continuous, non-negative variable representing the total amount paid by all parties for outpatient prescription medications as reported in Part D claims during the baseline period. |
| OOP pharmacy spending | A continuous, non-negative variable representing the total amount paid out-of-pocket by the beneficiary for outpatient prescription medications as reported in Part D claims during the baseline period. |
| Inpatient hospitalization use and | spending |
| Any inpatient stay | A binary indicator for whether a beneficiary had at least one inpatient hospitalization for any cause during the baseline period. |
| Inpatient stay count | A count of the number of inpatient hospitalizations for any cause a beneficiary had during the baseline period. |
| Inpatient length of stay | A count of the number of days (length of stay) a beneficiary was hospitalized in an inpatient facility during the baseline period. Length of stay for each inpatient hospitalization claim will be calculated as the arithmetic difference between each claim's from and through dates. |
| Total inpatient spending | A continuous, non-negative variable representing the total amount paid by all parties for all inpatient |

| Variable | Description |
|---|---|
| | hospitalizations (for any cause) as reported in inpatient facility claims during the baseline period. This is calculated as the sum of the Medicare payment amount, the Medicare per diem amount, the non-Medicare payer amount, and the patient OOP amount. |
| OOP inpatient spending | A continuous, non-negative variable representing the total amount paid out-of-pocket by the beneficiary for all inpatient hospitalizations (for any cause) as reported in inpatient facility claims during the baseline period. |
| Outpatient facility use and spending | |
| Any outpatient visit | A binary indicator for whether a beneficiary had at least<br>one claim for services provided by an outpatient facility<br>for any cause during the baseline period. |
| Outpatient visit count | A count of the number of unique dates with an outpatient facility for any cause claim a beneficiary had during the baseline period. |
| Total outpatient spending | A continuous, non-negative variable representing the total amount paid by all parties for outpatient facility claims during the baseline period. This is calculated as the sum of the Medicare payment amount, the blood deductible liability amount, the non-Medicare payer amount, and the patient OOP amount. |
| OOP outpatient spending | A continuous, non-negative variable representing the total amount paid out-of-pocket by the beneficiary for services as reported in outpatient facility claims during the baseline period. |
| Home health use and spending | |
| Any home health | A binary indicator for whether a beneficiary had at least<br>one claim for home health services during the baseline<br>period. |
| Home health count | A count of the number of home health visits a beneficiary had during the baseline period, calculated by summing the total visit count on each claim across claims. |
| Total home health spending | A continuous, non-negative variable representing the total amount paid by all parties for home health claims during the baseline period. This is calculated as the sum of the Medicare payment amount, the blood deductible liability amount, the non-Medicare payer amount, and the patient OOP amount. |

| Variable | Description |
|---|---|
| Part B spending | |
| Total Part B spending | A continuous, non-negative variable representing the total amount paid by all parties for Carrier and Durable Medical Equipment claims during the baseline period, calculated as the sum of the allowed amounts on each claim. |
| OOP Part B spending | A continuous, non-negative variable representing the total amount paid out-of-pocket by the beneficiary for Carrier and Durable Medical Equipment claims during the baseline period. |
| Total spending | |
| Total medical spending | A continuous non-negative variable representing the total amount paid by all parties for all medical services during the baseline period, including inpatient, outpatient, home health and Part B. |
| Total spending | A continuous non-negative variable representing the total amount paid by all parties for all medical and pharmacy claims during the baseline period and will be calculated as the sum of total pharmacy and total medical spending. |
| Other use | |
| Any ED visit | A binary indicator for whether a beneficiary had at least one emergency department visit during the baseline visit. Note that hospitals bill for emergency department visits on either the Inpatient or Outpatient facility claims, as described by there. Thus, emergency department visits will be identified in inpatient and outpatient facility claims via the presence of revenue center codes and . |
| ED visit count | A count of the number of unique dates with an emergency department visit that a beneficiary had during the baseline period. |
| Any pulmonology visit | A binary indicator for whether a beneficiary was treated<br>by a specialist in pulmonary disease during the baseline<br>period. Treatment by a pulmonologist will be identified<br>by the presence of a pulmonary specialty code in<br>inpatient, outpatient and Carrier claims. |
| Pulmonology visit count | A count of the number of unique dates with treatment<br>by a specialist in pulmonary disease that a beneficiary<br>had during the baseline period. |

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Variable | Description |
|---|---|
| Pulmonology prescriber | A binary indicator for whether the clinician who prescribed the beneficiary's index nintedanib medication was a pulmonologist, as documented in the Part D Prescriber Characteristics file for the index nintedanib claim. |

#### **Inflation Adjustment**

All dollar-denominated variables will be inflated to 2019 USD using the Consumer Price Index, which is listed in <u>Table 1</u>.

Table 1 Consumer price index for medical care implicit price deflator

| Year | Inflation Multiplier |
|------|----------------------|
| 2013 | 1.180 |
| 2014 | 1.152 |
| 2015 | 1.123 |
| 2016 | 1.077 |
| 2017 | 1.057 |
| 2018 | 1.038 |
| 2019 | 1.000 |

Source: U.S. BUREAU OF LABOR STATISTICS; Bureau of Labor Statistics Data (bls.gov), July 22, 2021.

#### 9.4 DATA SOURCES

As described above in <u>Section 9.2.1</u>, all variables will be constructed from the 100% Medicare claims and enrolment data from the U.S. Medicare program for the individuals meeting the sample selection criteria. To allow for a one-year baseline period and one-year follow-up period for all beneficiaries who initiated nintedanib between 10/01/2014 and 12/31/2018, the Medicare will span 10/01/2013 through 12/31/2019.

#### 9.5 STUDY SIZE

This study will use the GBTM technique to adherence pattern. Based on empirical results generated by resampling of population data, the maximum likelihood estimates obtained in group-based trajectory models provide reasonably close estimates of their true population values and have approximately normal distributions, even when estimated with a sample size as small as n = 500 (Loughran and Nagin, 2006). A prior study found 1,464 Medicare

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

beneficiaries who initiated nintedanib between 10/15/2014 and 12/31/2015 (<u>Corral, Chang et al., 2020</u>). By covering a longer period with the same data, this study should have a sufficient sample.

#### 9.6 DATA MANAGEMENT

| Pursuant to requirements guiding participation in the Innovator program, staff will access the Medicare claims and enrolment data only through the As such, will not directly possess any beneficiary-level data, and the only data to be downloaded from the summary-level statistics. |
|---|
| staff will access the environment via the VMware Horizon Client (or whichever client is mandated by from dedicated computers. All computers are secured with Microsoft BitLocker (for hard drive encryption at rest), Microsoft Azure Active Directory (to implement local security policies, including password management), BitDefender (anti-virus software), and LoJack (for computer tracking and remote wiping if ever needed). |
| All data manipulation and analysis will be conducted on the remotely by staff. Data manipulation and analysis will be conducted using SAS software ( ) and Stata software ( ). |

#### 9.7 DATA ANALYSIS

## 9.7.1 Main analysis

The objective of the main analysis is to identify the adherence patterns of nintedanib among IPF patients. The unit of analysis will be the individual beneficiary, each of whom will have twelve 30-days time intervals measurments of nintedanib PDC spanning the follow-up period. The 12 PDC values (PDC01–PDC12) will be characterized descriptively with measured of central tendency (mean, median), spread (min, max, interquartile range), and proportions of beneficiaries with PDC in each of 0 to <20%, 20 to <40%, 40 to <60%, 60 to <80%, and 80 to 100%.

GBTM will be used to explore the presence of distinct trajectories based on the change in medication adherence over time. The output of GBTM will include estimated probabilities of cluster membership for each individual and an estimated trajectory curve over time for each cluster. Different models will be used to identify 2 to 5 groups by using either cubic, quadratic, or quartic terms. The final models will be based on Bayesian information criteria, and Nagin's criteria for model adequacy (Nagin and Odgers, 2010), with consideration given to group size such that the proportion of patients in each group is not less than 5% of the total sample. The output of the final model will give us the estimated average trajectory for each group, as well as the estimated probabilities of membership in each trajectory for each patient. We will decide the number and shapes of trajectories based on both model fit,

ensuring enough class size and clinical usefulness (<u>Hickson, et al, 2020</u>). An example of using GBTM for assessing medication adherence is provided in Figure 2.



Figure 2 GBTM medication adherence example

Two sensitivity analyses will be conducted:

- First, the analysis will be repeated for beneficiaries who have positive PDC in the fourth month. In these models, only data from months 4 through 12 will be used to estimate the GBTMs because PDC01–PDC03 will have been used to condition the estimation sample.
- Second, the GBTMs will be re-estimated using as the outcome continuous PDC (for the same twelve30-day time intervals) and the beta distribution (Elmer, Jones and Nagin, 2018).

For each trajectory group identified, the mean PDC and the percent of beneficiaries in that group who discontinued nintedanib will be calculated.

## 9.7.2 Additional analysis

The objective of the additional analysis is to understand characteristics of patients within each nintedanib adherence trajectory among IPF patients. The unit of analysis will be the individual beneficiary, and the outcomes will be the vector of estimated probabilities of

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

cluster membership from a given GBTM. The predictor variables will be the baseline covariates (Section 9.3.3).

The distributions of the covariates will be characterized with descriptive statistics, including frequencies and percentages for discrete or categorical variables, and means, standard deviations, medians, and interquartile ranges for continuous variables.

Associations between the predictors and the probabilities of trajectory membership will be quantified using fractional multinomial logit models estimated via quasi-maximum likelihood (Papke and Wooldridge, 1996). Associations will be calculated both as odds ratios (exponentating the fractional multinomial logit model's coefficients) and average marginal effects on the probability scale.

## 9.8 QUALITY CONTROL

| The Medicare administrative data collection occurred in the past and the data will be obtained from . No additional insight into the data collection procedures is available beyond that which has been published by . As a result, we are relying on quality control measures implemented by . during data collection. |
|---|
| has established protocols for quality control of analyses. All analyses are audited before the finalization of results. The auditor will independently review the conceptual and technical elements of the analysis with a critical eye to identifying any flaws or potential errors. |

The auditor will understand the goal of the analysis and the expected results, and then review each step of the data analysis audit checklist (available upon request). The auditor will keep a list of questions or issues and then meet with the project lead to discuss any findings. If errors or issues are found that change the results, the auditor will perform an incremental audit to ensure that changes have been implemented properly and any change in results aligns with expectations about magnitude and direction.

#### 9.9 LIMITATIONS OF THE RESEARCH METHODS

This study has several limitations, which include:

- Absence of data on some behavioral factors (e.g. patient-physician communication, fear of disease/side effects, and family support) which may affect non-adherence.
- Reliance on prescription fill data to define adherence may not capture the actual use of the medication.
- In this study, patients who had 12 months of continued fee-for-service enrollment of Parts A, B, and D before and after index dates were included.

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 9.10 OTHER ASPECTS

#### 9.10.1 Data quality assurance

The following quality assurance and quality control measures will be applied to all programming that executes data extraction and transformation by

- Check program logs for notes, warning messages, and errors
- Check derived data values against source data for a patient sample to ensure correct derivation
- Verify that variables needed to support tables/listings/figures/ are found in the derived data set
- Check that data fields are not truncated
- Check data points for values outside expected ranges, where appropriate
- Check that data are rounded correctly and in accordance to the analysis plan
- Check that abbreviations, range categories, and subgroups conform to the analysis plan
- Ensure the consistency of sample counts across relevant tables/listings/figures
- Check formats consistent with the analysis plan
- Ensure no typos, misspellings, or false values
- Check that summary statistics are correct; check at least one category in each summary table against the data listings
- Check that data are in accordance with the Data Plan
- Check that subgroups conform to the Data Plan
- Ensure there are no duplicate observations

#### 9.10.2 Study records

Not applicable

# 10. PROTECTION OF HUMAN SUBJECTS

Not applicable based on secondary use of data without access to identifiable patient data.

# 10.1 STUDY APPROVAL, PATIENT INFORMATION, AND INFORMED CONSENT

Not applicable to this study.

## 10.2 STATEMENT OF CONFIDENTIALITY

Not applicable to this study

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 11. MANAGEMENT AND REPORTING OF ADVERSE EVENTS/ADVERSE REACTIONS

Given the information available within the Medicare claims database for this study, extraction on adverse events data will not be conducted and only data related to the study objectives will be extracted. Therefore, information about individual adverse events will not be available. Only data on aggregate-level medication use will be analysed.

# 11.1 ADVERSE EVENT AND SERIOUS ADVERSE EVENT COLLECTION AND REPORTING

Not applicable based on secondary use of data without any potential that any employee of BI or will access individually identifiable patient data.

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 12. PLANS FOR DISSEMINATING AND COMMUNICATING STUDY RESULTS

The results of this study will be considered for dissemination in the form of scientific publications (e.g., an abstract/poster for presentation at a national conference, a manuscript for submission to a peer-reviewed journal).

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 13. REFERENCES

#### 13.1 PUBLISHED REFERENCES

Alhazami M, Pontinha VM, Patterson JA, Holdford DA. Medication adherence trajectories: a systematic literature review. Journal of Managed Care & Specialty Pharmacy. 2020 Sep;26(9):1138-52.

Bateman BT, Franklin JM, Bykov K, Avorn J, Shrank WH, Brennan TA, Landon JE, Rathmell JP, Huybrechts KF, Fischer MA, Choudhry NK. Persistent opioid use following cesarean delivery: patterns and predictors among opioid-naive women. American journal of obstetrics and gynecology. 2016 Sep 1;215(3):353-e1.

Butler DC, Petterson S, Phillips RL, Bazemore AW. Measures of social deprivation that predict health care access and need within a rational area of primary care service delivery. Health services research. 2013 Apr;48(2pt1):539-59.

Cancer Medications Enquiry Database (CanMED). Surveillance Research Program SEER website tool. Division of Cancer Control and Population Sciences, National Cancer Institute. Version 1.9.1, 2021. Available at https://seer.cancer.gov/oncologytoolbox/canmed/. Accessed on May 27, 2021.

Corral M, Chang E, Broder MS, Gokhale S, Reddy SR. Healthcare use and costs among Medicare enrollees on pirfenidone versus nintedanib for idiopathic pulmonary fibrosis. Journal of Comparative Effectiveness Research. 2020 Jul;9(13):933-43.

Corral M, DeYoung K, Kong AM. Treatment patterns, healthcare resource utilization, and costs among patients with idiopathic pulmonary fibrosis treated with antifibrotic medications in US-based commercial and Medicare Supplemental claims databases: a retrospective cohort study. BMC Pulmonary Medicine. 2020 Dec;20(1):1-2.

Cutler RL, Fernandez-Llimos F, Frommer M, Benrimoj C, Garcia-Cardenas V. Economic impact of medication non-adherence by disease groups: a systematic review. BMJ open. 2018 Jan 1;8(1):e016982.

Desai R, Thakkar S, Fong HK, Varma Y, Khan MZ, Itare VB, Raina JS, Savani S, Damarlapally N, Doshi RP, Gangani K. Rising trends in medication non-compliance and associated worsening cardiovascular and cerebrovascular outcomes among hospitalized adults across the United States. Cureus. 2019 Aug;11(8).

Dillon P, Stewart D, Smith SM, Gallagher P, Cousins G. Group-based trajectory models: assessing adherence to antihypertensive medication in older adults in a community pharmacy setting. Clinical Pharmacology & Therapeutics. 2018 Jun;103(6):1052-60.

Dunn A, Grosse SD, Zuvekas SH. Adjusting health expenditures for inflation: a review of measures for health services research in the United States. Health Services Research. 2018 Feb;53(1):175-96.

Elmer J, Jones BL, Nagin DS. Using the Beta distribution in group-based trajectory models. BMC medical research methodology. 2018 Dec;18(1):1-5.

Farmer KC. Methods for measuring and monitoring medication regimen adherence in clinical trials and clinical practice. Clinical therapeutics. 1999 Jun 1;21(6):1074-90.

Feldman CH, Collins J, Zhang Z, Subramanian SV, Solomon DH, Kawachi I, Costenbader KH. Dynamic patterns and predictors of hydroxychloroquine nonadherence among Medicaid beneficiaries with systemic lupus erythematosus. In: Seminars in arthritis and rheumatism 2018 Oct 1 (Vol. 48, No. 2, pp. 205-213). WB Saunders.

Franklin JM, Gopalakrishnan C, Krumme AA, Singh K, Rogers JR, Kimura J, McKay C, McElwee NE, Choudhry NK. The relative benefits of claims and electronic health record data for predicting medication adherence trajectory. American heart journal. 2018 Mar 1;197:153-62.

Franklin JM, Krumme AA, Shrank WH, Matlin OS, Brennan TA, Choudhry NK. Predicting adherence trajectory using initial patterns of medication filling. Am J Manag Care. 2015 Sep 1;21(9):e537-44.

Franklin JM, Shrank WH, Pakes J, Sanfélix-Gimeno G, Matlin OS, Brennan TA, Choudhry NK. Group-based trajectory models: a new approach to classifying and predicting long-term medication adherence. Medical care. 2013 Sep 1:789-96.

Forbes CA, Deshpande S, Sorio-Vilela F, Kutikova L, Duffy S, Gouni-Berthold I, Hagström E. A systematic literature review comparing methods for the measurement of patient persistence and adherence. Current medical research and opinion. 2018 Sep 2;34(9):1613-25.

Gagne JJ, Glynn RJ, Avorn J, Levin R, Schneeweiss S. A combined comorbidity score predicted mortality in elderly patients better than existing scores. Journal of clinical epidemiology. 2011 Jul 1:64(7):749-59.

Harbaugh CM, Cooper JN. Administrative databases. InSeminars in pediatric surgery 2018 Dec 1 (Vol. 27, No. 6, pp. 353-360). WB Saunders.

Hargrove JL, Pate V, Casteel CH, Golightly YM, Loehr LR, Marshall SW, Stürmer T. Antihypertensive adherence trajectories among older adults in the first year after initiation of therapy. American journal of hypertension. 2017 Oct 1;30(10):1015-23.

Hickson, R.P., et al., Opening the black box of the group-based trajectory modeling process to analyze medication adherence patterns: An example using real-world statin adherence data. Pharmacoepidemiology and drug safety, 2020. 29(3): p. 357-362.

Ipatova AY, Koerner PH, Miller RT, Staskon F, Radi M. Retrospective analysis of medication utilization and clinical outcomes in patients with idiopathic pulmonary fibrosis treated with nintedanib or pirfenidone. Clinical Medicine Insights: Circulatory, Respiratory and Pulmonary Medicine. 2019 Mar;13:1179548419834922.

Jones BL, Nagin DS. A note on a Stata plugin for estimating group-based trajectory models. Sociological Methods & Research. 2013 Nov;42(4):608-13.

Juarez DT, Williams AE, Chen C, Daida YG, Tanaka SK, Trinacty CM, Vogt TM. Factors affecting medication adherence trajectories for patients with heart failure. The American journal of managed care. 2015 Mar 1;21(3):e197.

Kim SC, Choudhry N, Franklin JM, Bykov K, Eikermann M, Lii J, Fischer MA, Bateman BT. Patterns and predictors of persistent opioid use following hip or knee arthroplasty. Osteoarthritis and cartilage. 2017 Sep 1;25(9):1399-406.

Lam WY, Fresco P. Medication adherence measures: an overview. BioMed research international. 2015 Oct 11;2015.

Li Y, Zhou H, Cai B, Kahler KH, Tian H, Gabriel S, Arcona S. Group-based trajectory modeling to assess adherence to biologics among patients with psoriasis. ClinicoEconomics and outcomes research: CEOR. 2014;6:197.

Lo-Ciganic WH, Gellad WF, Gordon AJ, Cochran G, Zemaitis MA, Cathers T, Kelley D, Donohue JM. Association between trajectories of buprenorphine treatment and emergency department and in-patient utilization. Addiction. 2016 May;111(5):892-902.

Loughran T, Nagin DS. Finite sample effects in group-based trajectory models. Sociological methods & research. 2006 Nov;35(2):250-78.

MacEwan JP, Forma FM, Shafrin J, Hatch A, Lakdawalla DN, Lindenmayer JP. Patterns of adherence to oral atypical antipsychotics among patients diagnosed with schizophrenia. Journal of managed care & specialty pharmacy. 2016 Nov;22(11):1349-61.

Nagin DS, Odgers CL. Group-based trajectory modeling in clinical research. Annual review of clinical psychology. 2010 Apr 27;6:109-38.

Papke LE, Wooldridge JM. Econometric methods for fractional response variables with an application to 401 (k) plan participation rates. Journal of applied econometrics. 1996 Nov;11(6):619-32.

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Paranjpe R, Johnson ML, Essien EJ, Barner JC, Serna O, Gallardo E, Majd Z, Fleming ML, Ordonez N, Holstad MM, Abughosh SM. Group-Based Trajectory Modeling to Identify Patterns of Adherence and Its Predictors Among Older Adults on Angiotensin-Converting Enzyme Inhibitors (ACEIs)/Angiotensin Receptor Blockers (ARBs). Patient preference and adherence. 2020;14:1935.

Raebel MA, Schmittdiel J, Karter AJ, Konieczny JL, Steiner JF. Standardizing terminology and definitions of medication adherence and persistence in research employing electronic databases. Medical care. 2013 Aug;51(8 0 3):S11.

Sun JW, Rogers JR, Her Q, Welch EC, Panozzo CA, Toh S, Gagne JJ. Adaptation and validation of the combined comorbidity score for ICD-10-CM. Medical care. 2017 Dec 1;55(12):1046-51.

Vadhariya A, Fleming ML, Johnson ML, Essien EJ, Serna O, Esse T, Choi J, Boklage SH, Abughosh SM. Group-based trajectory models to identify sociodemographic and clinical predictors of adherence patterns to statin therapy among older adults. American health & drug benefits. 2019 Jun;12(4):202.

Wang X, Chen H, Essien E, Wu J, Serna O, Paranjpe R, Abughosh S. Medication adherence to antihypertensive triple-combination therapy among patients enrolled in a medicare advantage plan. Journal of managed care & specialty pharmacy. 2019 Jun;25(6):678-86.

Zongo A, Simpson S, Johnson JA, Eurich DT. Change in Trajectories of Adherence to Lipid-Lowering Drugs Following Non-Fatal Acute Coronary Syndrome or Stroke. Journal of the American Heart Association. 2019 Dec 3;8(23):e013857.

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 14. ANNEXURES

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## ANNEX 1. LIST OF STAND-ALONE DOCUMENTS

| Number | Document<br>Reference Number | Date | Title |
|--------|------------------------------|-------------|----------------|
| 1 | <number></number> | July 7 2021 | Code_List.xlsx |

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### ANNEX 2. ENCEPP CHECKLIST FOR STUDY PROTOCOLS

A copy of the European Network of Centers for Pharmacoepidemiology and Pharmacovigilance (ENCePP) Checklist for Study protocols available at website: encepp.eu/standards\_and\_guidances/index.html completed and signed by the main author of the study protocol should be included in Annex 2.

The checklist will facilitate the review of the protocol and evaluation of whether investigators have considered important methodological aspects.

In question 9.5 of the Checklist, Revision 1:

- "Study start" means "Start of data collection"
- "Study progress" means "Progress report(s)"
- "Study completion" means "End of data collection"
- "Reporting" means "Final report of the study results"

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## **ANNEX 3. ADDITIONAL INFORMATION**

Additional annexes may be included if necessary.

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## ANNEX 4. REVIEWERS AND APPROVAL SIGNATURES

The NIS Protocol must be sent for review to the following individuals prior to approval.

| Reviewer | NIS involving BI product(s) | NIS not invo | lving BI product(s) |
|---|---|---|---|
| | | Global NIS | Local NIS |
| NIS Lead | X | X | X |
| Global TM Epi | X | X | X |
| Global TMM / TMMA / TM Market<br>Access | X | X | |
| Global Project Statistician | X | X | |
| Global TM RA | X | | |
| Global PVWG Chair | X | | |
| GPV SC | X | X | X |
| Global CTIS representative | X | | |
| Local Medical Director | X (if local study) | | X |
| Local Head MAcc / HEOR Director | X (if local study) | | X |
| Global TA Head Epi* | X | X | |
| Global TA Head Clinical Development / Medical Affairs / Market Access* | X | X | |
| Global TA Head PV RM* | X | | |
| RWE CoE | X | X | |
| PSTAT / PSTAT-MA<br>(for NISnd only) | X | X | X |
| NIS DM | X | X | X |
| Local Head MA/Clinical Development | | | X (does not apply to<br>NISed without chart<br>abstraction) |

<sup>\*</sup> After review by Global TM for function

Include this Annex if signatures of external investigators are required and/or for studies that will not be stored in the DMS for submission documents. For non-interventional studies approval signatures must be obtained from the individuals as noted in section 5.1.3 "Manage NIS Protocol" in the corresponding SOP 001-MCS-90-118. If the study is a PASS, additional approvals are necessary; refer to SOP 001-MCS-90-140 "Post Authorization Safety Studies".

# Non-Interventional Study (NIS) Protocol

# **BI Study Number 1199-0471**

c39084239-01

| Study Title: Study Number: Protocol Version: I herewith certify that I agree to the content of the study protocol and to all documents referenced in the study protocol. Note: Please insert respective signatories with regard to the SOP. | | |
|---|---|---|
| Position: NIS Lead | Name/Date: <> | Signature: |
| Position: | Name/Date: | Signature: |
| Position: | Name/Date: | Signature: |
| Position: | Name/Date: | Signature: |
| Position: | Name/Date: | Signature: |
| Position: | Name/Date: | Signature: |